CLINICAL TRIAL: NCT05558371
Title: Multi-Site Validation of Biomarkers and Core Clinical Outcome Measures for Clinical Trials Readiness in CDKL5 Deficiency Disorder
Brief Title: International CDKL5 Clinical Research Network
Acronym: ICCRN
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); International Foundation for CDKL5 Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-2756; 5U01NS114312 (NIH)
Record Dates: First submitted 2022-07-28; First posted 2022-09-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: CDKL5; CDKL5 Deficiency Disorder; CDD
MeSH Terms: conditions — CDKL5 deficiency disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. — No intervention administered as part of this study; observational only.

SUMMARY:
Pathogenic variants in the Cyclin-dependent kinase like 5 (CDKL5) gene cause CDKL5 deficiency disorder (CDD, MIM 300672, 105830), a severe developmental and epileptic encephalopathy associated with cognitive and motor impairments and cortical visual impairment. While capability for disease modifying therapies is accelerating, there is a critical barrier for clinical trial readiness that may result in failure of these therapies, not due to lack of efficacy but due to lack of validated outcome measures and biomarkers. The measures and biomarkers validated here will be adaptable to other developmental and epileptic encephalopathies.

DETAILED DESCRIPTION:
Pathogenic variants in the Cyclin-dependent kinase like 5 (CDKL5) gene cause CDKL5 deficiency disorder (CDD, MIM 300672, 105830) a severe developmental and epileptic encephalopathy (DEE) associated with cognitive and motor dysfunction and cortical visual impairment. Recent data suggest CDD is one of the most common genetic causes of DEE. Work in CDD animal models has demonstrated the ability for disease modification and symptom reversal: worldwide efforts are now underway to develop therapeutic strategies (including gene therapy) to treat and potentially cure CDD. While there are four active clinical trials, none assesses the full spectrum of this DEE to address true disease modification. While capability for disease modifying therapies is accelerating, there is a critical barrier for clinical trial readiness that may result in failure of these therapies, not due to lack of efficacy but due to lack of validated outcome measures.

CDD has been associated historically with Rett syndrome but there are many clear distinctions and CDD has emerged as an independent disorder. Some Clinical Outcome Measures (COMs) can be adapted from Rett syndrome COMs, whereas others need to be developed specifically for CDD. Our research network is uniquely positioned to develop clinical trial readiness for CDD by pairing exceptional experience in the development and validation of outcome measures with an extensive network of CDD experts and clinical trialists. Our goals are to 1) refine and validate appropriate quantitative COMs and biomarkers and 2) conduct a multi-site clinical trial readiness study to ensure that they can be successfully implemented. We will test the hypothesis that CDD specific COMs can be refined to accurately and reproducibly track meaningful changes in clinical trials:

Aim 1: Generate and validate a suite of COMs and biomarkers necessary to comprehensively assess disease modification in CDD.

Aim 2: Conduct a multi-site clinical trial readiness study to assess implementation, longitudinal stability, and collect baseline COMs and EEG/evoked potential data.

Overall Impact: These outcome measures will establish clinical trial readiness for CDD and generate historic baseline outcome data, ensuring optimal testing of potential new therapeutics including gene therapy. Furthermore, these measures will be adaptable to other DEEs by enabling choices of outcome measures beyond existing NINDS supported measurement tools (NeuroQoL, PROMIS, Toolbox) that are not designed for the severity of the DEE populations.

ELIGIBILITY:
Inclusion Criteria:

* All children diagnosed with CDD age 1-month to 100 years of age that are receiving care at one of the study institutions or are registered with the International CDKL5 Disorder Database will be considered for the study population.

Exclusion Criteria:

* Individuals who do not meet study inclusion criteria.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CDKL5 Deficiency Disorder (CDD).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
CDKL5 Deficiency Disorder (CDD) Clinical Severity Assessment - Clinician (CCSA-Clinician) | 5 years
  Measured by clinician rating of patient. Item scores are transformed to a scale of 0-100 and the total score is calculated as a mean item score. Higher scores indicate higher severity.
CDKL5 Deficiency Disorder (CDD) Clinical Severity Assessment - Caregiver (CCSA-Caregiver) | 5 years
  Measured by caregiver/parent rating of patient on a scale of 0-100 with a higher score indicating higher severity.
CDKL5 Deficiency Disorder (CDD) Development Questionnaire - Caregiver (CDQ-Caregiver) | 5 years
  Measured by caregiver/parent rating of patient on a scale of 0-100 with a higher score indicating higher severity.
Communication and Symbolic Behavior Scales - Developmental Profile Infant Toddler Checklist (CSBS-DP ITC) | 5 years
  Measured by caregiver/parent rating of patient on a 24-item questionnaire. Three composite scores and a total score can be derived. Items contribute to the 0-57 point scale for the total score with lower scores indicating concerns for communication skills.
Sleep Disorder Scale for Children (SDSC) | 5 years
  Measured by caregiver/parent rating of patient on a 26- Likert type item questionnaire. Scale goes from 0-39 with a higher score indicating higher severity of sleep disorder. Each subscale is scored through the summation of all the subscale items. Comparing scores were the normative data reported in the initial validation paper, z-scores and t-scores can be derived. The t-score enables scores to be dichotomized as within normal range or outside of normal range, compared to the general population.
Quality of Life Inventory - Disability (QI-Disability) | 5 years
  This is a quality of life measure for children with intellectual disability. The measure comprises 32 items that are rated on a five-point Likert scale and group into six subscales: physical health, positive emotions, negative emotions, social interactions, independence, and leisure and outdoors. Following transformation to a 100-point scale, item scores in each subscale are summed and divided by the number of items to give a subscale score. The mean of the six subscale scores is calculated to give the total QOL score.
CDKL5 Deficiency Disorder (CDD) Gross Motor (CDD-Motor) | 5 years
  This is a video measure of gross motor function, based on the Rett Syndrome Gross Motor Scale with additional items that enable measurement of head control and sitting. Parents are provided with a filming protocol, video clips are uploaded to the investigators, and data are coded according to a predetermined coding system.
CDKL5 Deficiency Disorder (CDD) Fine Motor (CDD-Hand) | 5 years
  This is a video measure of fine motor function based on the Rett Syndrome Hand Function Scale with additional instructions on filming for if the patient has Cortical Visual Impairment. Parents are provided with a filming protocol, video clips are uploaded to the investigators, and data are coded according to a predetermined coding system.
Electroencephalogram/Evoked Potentials (EEG/EP) characteristics in CDKL5 Deficiency Disorder. | 5 years
  Measured by correlations of EEG/EP with other study scales.

SECONDARY OUTCOMES:
Frequency of different mutations in the CDKL5 Deficiency Disorder population | 5 years
  Measured by information obtained from genetic reports of enrolled participants.
Frequency of medications and their indications in the CDKL5 Deficiency Disorder population | 5 years
  Measured by medication/indication data obtained from medical record review and/or caregiver report.
Social Determinants of Health (SDOH) in CDKL5 Deficiency Disorder population | 5 years
  Measured by data elements that are collected to describe the socioeconomic status of the study population. Examples include caregiver education level, marital status and employment status, patient living situation, household income, and primary caregiver information.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Benke, MD PhD, Principal Investigator — University of Colorado, Denver
Locations (9):
- United States (8):
  - University of California Los Angeles/UCLA Mattel Children's Hospital, Los Angeles, California
  - University of Colorado Denver/Children's Hospital Colorado, Aurora, Colorado
  - Harvard Medical School/Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis/St. Louis Children's Hospital, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/ Texas Children's Hospital, Houston, Texas
- Telethon Kids Institute/Perth Children's Hospital, Perth, Nedlands Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
The ICCRN will be utilizing the National Institute of Mental Health (NIMH) Data Archive (NDA), previously known as the National Database for Autism Research (NDAR), as our final deidentified repository of our data. We will utilize Global Unique Identifiers to ensure we have deconflicted patient data across all institutions. Each institution will be directly uploading patient data to our central REDCap database to allow for cleaning of data prior to upload to NDA. Our data elements will be harmonized with other NDA elements where appropriate at the start of the study. The one exception is patient videos which will be reviewed at Telethon kids secure network for analysis, but the scored results of validated motor scales will be uploaded to NDAR in a deidentified fashion. All scales, outcome measures, and protocols (both for scoring and implementation of COMs) will also be shared through publications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available data will be released to the repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first.
Access Criteria: NIMH NDA policy will govern access criteria.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Olson HE, Daniels CI, Haviland I, Swanson LC, Greene CA, Denny AMM, Demarest ST, Pestana-Knight E, Zhang X, Moosa AN, Fidell A, Weisenberg JL, Suter B, Fu C, Neul JL, Percy AK, Marsh ED, Benke TA, Poduri A. Current neurologic treatment and emerging therapies in CDKL5 deficiency disorder. J Neurodev Disord. 2021 Sep 16;13(1):40. doi: 10.1186/s11689-021-09384-z. PMID 34530725
- [Background] Brock D, Fidell A, Thomas J, Juarez-Colunga E, Benke TA, Demarest S. Cerebral Visual Impairment in CDKL5 Deficiency Disorder Correlates With Developmental Achievement. J Child Neurol. 2021 Oct;36(11):974-980. doi: 10.1177/08830738211019284. PMID 34547934
- [Background] Saldaris J, Weisenberg J, Pestana-Knight E, Marsh ED, Suter B, Rajaraman R, Heidary G, Olson HE, Devinsky O, Price D, Jacoby P, Leonard H, Benke TA, Demarest S, Downs J. Content Validation of Clinician-Reported Items for a Severity Measure for CDKL5 Deficiency Disorder. J Child Neurol. 2021 Oct;36(11):998-1006. doi: 10.1177/08830738211019576. Epub 2021 Aug 11. PMID 34378447
- [Background] Olson HE, Costantini JG, Swanson LC, Kaufmann WE, Benke TA, Fulton AB, Hansen R, Poduri A, Heidary G. Cerebral visual impairment in CDKL5 deficiency disorder: vision as an outcome measure. Dev Med Child Neurol. 2021 Nov;63(11):1308-1315. doi: 10.1111/dmcn.14908. Epub 2021 May 24. PMID 34028805
- [Background] MacKay CI, Bick D, Prokop JW, Munoz I, Rouse J, Downs J, Leonard H. Expanding the phenotype of the CDKL5 deficiency disorder: Are seizures mandatory? Am J Med Genet A. 2020 May;182(5):1217-1222. doi: 10.1002/ajmg.a.61504. Epub 2020 Feb 8. PMID 32034940
- [Background] Dale T, Downs J, Wong K, Leonard H. The perceived effects of cannabis products in the management of seizures in CDKL5 Deficiency Disorder. Epilepsy Behav. 2021 Sep;122:108152. doi: 10.1016/j.yebeh.2021.108152. Epub 2021 Jun 18. PMID 34148781
- [Background] Leonard H, Junaid M, Wong K, Demarest S, Downs J. Exploring quality of life in individuals with a severe developmental and epileptic encephalopathy, CDKL5 Deficiency Disorder. Epilepsy Res. 2021 Jan;169:106521. doi: 10.1016/j.eplepsyres.2020.106521. Epub 2020 Dec 1. PMID 33341033
- [Background] MacKay CI, Wong K, Demarest ST, Benke TA, Downs J, Leonard H. Exploring genotype-phenotype relationships in the CDKL5 deficiency disorder using an international dataset. Clin Genet. 2021 Jan;99(1):157-165. doi: 10.1111/cge.13862. Epub 2020 Oct 20. PMID 33047306
- [Background] Benke TA, Kind PC. Proof-of-concept for a gene replacement approach to CDKL5 deficiency disorder. Brain. 2020 Mar 1;143(3):716-718. doi: 10.1093/brain/awaa055. PMID 32203572